CLINICAL TRIAL: NCT05257863
Title: Development of Machine Learning Models for the Prediction of Complications After Colonic, Colorectal and Small Intestine Anastomosis in Psychiatric and Non-psychiatric Patient Collectives (P-Study)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr. Med Anas Taha (Other)
Collaborators: University of Basel (Other); University of Hamburg-Eppendorf (Other)
Responsible Party: Sponsor-Investigator, Dr. Med Anas Taha, Research Fellow, University of Basel
Organization: University of Basel (Other)
Other Study IDs: P-Study
Record Dates: First submitted 2022-01-21; First posted 2022-02-25 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Postoperative Complications; Psychosomatic Disorder; Psychiatric Disorder; Cancer; Diverticulitis; Morbus Crohn; Colitis Ulcerosa; Anastomotic Leak; Anastomotic Complication; Small Intestine Anastomotic Leak
Keywords: machine learning; clinical prediction modeling; artificial intelligence
MeSH Terms: conditions — Postoperative Complications; Psychophysiologic Disorders; Mental Disorders; Neoplasms; Diverticulitis; Crohn Disease; Colitis, Ulcerative; Anastomotic Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our study aims to lay the basis for a predictive modeling service for postoperative complications and prolonged hospital stay in patients suffering from psychiatric diseases undergoing colorectal surgery.

Furthermore, we aim to investigate the impact of preoperative Risk factors, psychiatric and psychosomatic diseases on the outcomes of colorectal surgery and the complications after colorectal surgeries like anastomosis insufficiency via predictive modeling techniques

The service mentioned above will be publicly available as a web-based application

ELIGIBILITY:
Inclusion Criteria:

* Colocolic, colorectal and small intestine anastomosis
* Neoplasia,
* Diverticulitis
* Mesenteric ischemia
* Iatrogenic or traumatic perforation
* Inflammatory bowel disease

Exclusion Criteria:

* Patients <18 years
* Patients suffering from recurrent colorectal cancer bearing
* Peritoneal carcinomatosis or unresectable metastatic disease at the time of bowel resection and anastomosis will be excluded.
* Patients who cannot be followed up on for more than six weeks after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing colorectal and small intestine surgery.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Anastomotic insufficiency/leakage | From index surgery up to six weeks postoperatively
  Predictive model with an app for the development of anastomosis insufficiency based on the risk factors.
Complication after surgery/ Comprehensive Complication Index/ Clavian Dindo Score | From index surgery up to six weeks postoperatively
  Impact of psychatric and psychosomatic disorders are having higher complication rates
Length of Hospital Stay (in Days) | From surgery up to 12 weeks postoperatively
  Impact of psychatric and psychosomatic disorders are having longer hospitalization
Intraoperative influid manangment | Time Frame: From index surgery up to six weeks postoperatively
  Impact of Intraoperative influid on the development of anastomotic insuffiency
Development of a preoperative score for morbidity/mortality in colorectal surgery | From index surgery up to six weeks postoperatively
  Check the risk for morbidity/mortality in colorectal surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University of Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided